CLINICAL TRIAL: NCT02130531
Title: Pharmacokinetic and Pharmacodynamic Study of Emixustat Hydrochloride in Subjects With Geographic Atrophy Associated With Dry Age-Related Macular Degeneration
Brief Title: Pharmacokinetic and Pharmacodynamic Study of Emixustat in Subjects With Geographic Atrophy Associated With Dry Age-Related Macular Degeneration
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kubota Vision Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 4429-101
Record Dates: First submitted 2014-05-01; First posted 2014-05-05 (Estimated); Last update posted 2016-01-18 (Estimated); Status verified 2016-01

CONDITIONS: Geographic Atrophy; Age-Related Macular Degeneration
MeSH Terms: conditions — Geographic Atrophy; Macular Degeneration | interventions — emixustat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort 1 (Experimental): Two dose periods in any sequence (subjects will be assigned to 1 of 2 possible sequences):
  * Emixustat HCl Tablet Strength B (mid dose); 1 tablet once daily & 1 placebo tablet once daily for 7 days
  * Emixustat HCl Tablet Strength A (low dose); 1 tablet twice daily for 7 days
  Interventions: Drug: Emixustat HCl Tablet; Other: Placebo Tablet
- Cohort 2 (Experimental): Three dose periods in any sequence (subjects will be assigned to 1 of 6 possible sequences):
  * Emixustat HCl Tablet Strength A (low dose); 1 tablet daily for 7 days
  * Emixustat HCl Tablet Strength B (mid dose); 1 tablet daily for 7 days
  * Emixustat HCl Tablet Strength C (high dose); 1 tablet daily for 7 days
  Interventions: Drug: Emixustat HCl Tablet

INTERVENTIONS:
Drug: Emixustat HCl Tablet — Tablet for oral administration
  Other Names: ACU-4429
Other: Placebo Tablet — Tablet for oral administration
  Arms: Cohort 1

SUMMARY:
The purpose of this study is to characterize emixustat hydrochloride pharmacokinetic and pharmacodynamic parameters in subjects with geographic atrophy associated with dry age-related macular degeneration.

DETAILED DESCRIPTION:
This is a multi-center, randomized, masked, multiple-dose, crossover study of the pharmacokinetics of emixustat hydrochloride (HCl) in subjects with geographic atrophy (GA) associated with dry age-related macular degeneration (AMD). Subjects will receive study drug during multiple dose periods in a crossover design, and serve as their own controls. There is a 21-28 day washout period between dose periods. The final Study Exit visit is 21 to 28 days after the subject's last dose of study drug at the end of the final dosing period.

ELIGIBILITY:
Inclusion Criteria:

* Males or females age ≥65 years
* Clinical diagnosis of GA associated with AMD
* Able and willing to provide written informed consent
* Able to reliably administer oral medication by self or with available assistance

Exclusion Criteria:

* Geographic atrophy associated with a condition other than AMD
* History of, active or high risk of developing choroidal neovascularization (CNV) in either eye
* Known serious allergy to the fluorescein sodium for injection in angiography
* Pre-specified laboratory abnormalities at screening
* Treatment with any investigational study drug within 30 days of screening or device within 60 days of screening
* Prior participation in any clinical study of emixustat
* History of other disease, metabolic dysfunction, chronic immunosuppression, physical examination finding
* Male subjects who are not surgically sterile and are not willing to practice a medically accepted method of birth control with their female partner of childbearing potential from screening through 21 days after the last dose of study drug

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 26 (Actual)
Dates: Start 2014-04; Primary Completion 2015-09 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Area Under the Concentration-Time Curve from time zero to 24 hours [(AUC(0-24h)] | Day 1 and Day 7 of each dosing period
Degree of suppression of the ERG b-wave response post-photobleaching. | Screening through Day 10 of each dosing period and study exit

CONTACTS AND LOCATIONS:
Overall Officials: Acucela Medical Monitor, Study Director — Kubota Vision Inc.
Locations (1):
- Call Acucela Clinical Trials Helpdesk for locations, Seattle, Washington, United States